CLINICAL TRIAL: NCT06456866
Title: Assessing the Accuracy of ChatGPT-4 in Interpreting Arterial Blood Gas Results
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, anesthesiology and reanimation specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: Blood gases
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Blood Gases
Keywords: artificial intelligence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ChatGPT
  Interventions: Other: interpretation
- Anesthesiology expert
  Interventions: Other: interpretation

INTERVENTIONS:
Other: interpretation — interpretation of blood gases samples

SUMMARY:
Assessment of Acidosis and Alkalosis, Evaluation of Hypoxemia and Hyperoxemia, Evaluation of Hemoglobin Parameters, Assessment of Electrolytes, Evaluation of Metabolic Parameters (Glucose, Lactate, Bilirubin)

DETAILED DESCRIPTION:
Model Training:

The collected data will be used to train the artificial intelligence model. Utilizing the deep learning infrastructure provided by ChatGPT Plus, our model will be optimized to produce highly accurate results in interpreting blood gases.

During the training process, our model will be taught to interpret various blood gas samples, including assessments of acidosis-alkalosis, hypoxemia-hyperoxemia, hemoglobin, electrolytes, and metabolic parameters.

Model Testing and Validation:

The trained model will be tested on previously unseen test datasets to evaluate its performance. This step is crucial for understanding how the model will perform in real-world scenarios.

The accuracy of the model will be assessed by comparing its interpretations with feedback provided by expert anesthesiologists.

Furthermore, to comprehensively evaluate ChatGPT's effectiveness in this domain, the daily arterial blood gas results obtained in the intensive care unit will be submitted to ChatGPT for interpretation. The same questions will be posed, and the responses will be evaluated by an anesthesiology and reanimation specialist. These questions will be asked to the model:

Assessment of Acidosis and Alkalosis, Evaluation of Hypoxemia and Hyperoxemia, Evaluation of Hemoglobin Parameters, Assessment of Electrolytes, Evaluation of Metabolic Parameters (Glucose, Lactate, Bilirubin)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and above will be included in the study.
* The study will evaluate arterial blood gas results.

Exclusion Criteria:

* Venous blood gas results,
* Blood gas results with calibration errors,
* Blood gas results with incomplete data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of 398 arterial blood gas samples from patients in the intensive care unit will be included in the study
Sampling Method: Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
blood gases sample interpretation | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
there will be no IPD in this research. The investigators will only use blood gases samples and delete all the IPD.